CLINICAL TRIAL: NCT04052282
Title: Test-retest Reliability and Validity of and a Novel Smartphone Application to Objectively Measure Physical Function in Healthy Individuals
Brief Title: A Novel Smartphone Application for "Smart" Trials
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Tufts Medical Center (Other)
Responsible Party: Principal Investigator, Lucas Ogura Dantas, Co-Principal Investigator, Universidade Federal de Sao Carlos
Other Study IDs: IRB #:13237
Record Dates: First submitted 2019-08-05; First posted 2019-08-09 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Technology; Physical Function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mobile Health App - Healthy Individuals: Mobile health App - Test
  Beta Testing 1: The Beta test 1 will be performed with participants inside the Research Center. The purpose of this phase is to increase usability, acceptability and reliability of the mHealth App in participants.
  Beta Testing 2: The Beta test 2 will be performed with patients outside the Research Center, at their houses. The purpose is to focus on the mHealth App remote usability, acceptability, and data collection.
  Interventions: Device: Mobile Health App

INTERVENTIONS:
Device: Mobile Health App — There is no intervention

SUMMARY:
The overarching goal is to develop a mHealth App that can use smartphone embedded sensors to objectively collect physical function data in healthy individuals in the context of daily life.

DETAILED DESCRIPTION:
The goal is to develop a mHealth App using smartphone embedded sensors to objectively collect physical function data in healthy individuals in the context of daily life. The investigators will perform technical development of an internet-interactive App to collect, analyze and transfer the subjects' data. As a proof-of-concept, the mHealth App will execute algorithms that automate deployment of three well-established physical function tests. In a laboratory setting, it will be evaluated usability, acceptability and reliability of the mHealth App compared with traditional performance tests among focus groups. The investigators will then evaluate its usability and acceptability when used in the participants' home environments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 50 years old with symptomatic knee osteoarthritis
* English Speaker
* Be able to walk 20 meters without an assistive device, such as a cane, walker or crutches.
* Have an iPhone 6 or higher with internet connection.

Exclusion Criteria:

* Prior surgery on either knee within 6 months of enrollment
* Received corticosteroid injection in the knee within 3 months of enrollment
* Evidence or history of knee disease or trauma

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes healthy subjects who are equal or greater than 50 years old.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale - TEST RETEST (clinical setting) | Day 1
  A Numeric Rating Scale (NRS) will be applied to measure both knee pain. NRS is a well recognized tool to measure the intensity of pain that visually represents the intensity of pain that the individual believes to present. The scale will be displayed on the app and will have a range of 0 to 10, with 0 being the complete absence of pain and 10, the maximum intensity of pain reported by the individual.
Numeric Rating Scale - TEST RETEST (clinical setting) | 7 days after day 1
  A Numeric Rating Scale (NRS) will be applied to measure both knee pain. NRS is a well recognized tool to measure the intensity of pain that visually represents the intensity of pain that the individual believes to present. The scale will be displayed on the app and will have a range of 0 to 10, with 0 being the complete absence of pain and 10, the maximum intensity of pain reported by the individual.
Numeric Rating Scale - DIURNAL CHANGE (home setting) | Day 1, day 3, and day 5 (within a week Mon, Wed, Fri)
  At home, a Numeric Rating Scale (NRS) will be applied to measure both knee pain. NRS is a well recognized tool to measure the intensity of pain that visually represents the intensity of pain that the individual believes to present. The scale will be displayed on the app and will have a range of 0 to 10, with 0 being the complete absence of pain and 10, the maximum intensity of pain reported by the individual.
The Get up and Go - TEST RETEST (clinical setting) | Day 1
  In the clinical setting, the clinician asks the patient to stand up from a chair, walk 3 meters, turn around, return and sit back in the chair. The time on the test is used as a predictor of functional independence: below 20 seconds is considered normal and over 30 seconds as potentially indicative of increased risk for falls and functional dependence. For the automated test, the patient will wear a chest strap fixing the mobile phone over the sternum. On a sitting position, the patient will open the mHealth App and through the use of audible feedback, will receive the same test instructions as in the clinic. With the use of algorithms, the mHealth App will pre-determine and tell the patient how many steps to take to achieve the distance of 3 meters. After the test is completed, the data will be automatically sent to the cloud system.
The Get up and Go - TEST RETEST (clinical setting) | 7 days after day 1
  In the clinical setting, the clinician asks the patient to stand up from a chair, walk 3 meters, turn around, return and sit back in the chair. The time on the test is used as a predictor of functional independence: below 20 seconds is considered normal and over 30 seconds as potentially indicative of increased risk for falls and functional dependence. For the automated test, the patient will wear a chest strap fixing the mobile phone over the sternum. On a sitting position, the patient will open the mHealth App and through the use of audible feedback, will receive the same test instructions as in the clinic. With the use of algorithms, the mHealth App will pre-determine and tell the patient how many steps to take to achieve the distance of 3 meters. After the test is completed, the data will be automatically sent to the cloud system.
The Get up and Go - DIURNAL CHANGE (home setting) | Day 1, day 3, and day 5 (within a week Mon, Wed, Fri)
  At home, for the automated test, the patient will wear a chest strap fixing the mobile phone over the sternum. On a sitting position, the patient will open the mHealth App and through the use of audible feedback, will receive the same test instructions as in the clinic. With the use of algorithms, the mHealth App will pre-determine and tell the patient how many steps to take to achieve the distance of 3 meters. After the test is completed, the data will be automatically sent to the cloud system.
The 30 Seconds Sit to Stand - TEST RETEST (clinical setting) | Day 1
  In the clinical setting, the clinician asks the patient to sit in the middle of the chair, with the back straight, feet apart resting on the floor and in line with the shoulders. The patient has to rise from a sitting to a standing position as many times as possible in 30 seconds. With the results of this test, it is possible to evaluate a wide variety of skill levels, with scores ranging from 0 (for those unable to complete one repetition) to more than 20 repetitions (for the most physically fit individuals). For the automated test, the patient will wear a chest strap fixing the mobile phone over the sternum. On a sitting position, the patient will open the mHealth App and through the use of audible feedback, will receive the same test instructions as in the clinic. With the use of algorithms, the mHealth App will automatically count the total sit to stand repetitions within a 30 seconds period. After the test is completed, the data will be automatically sent to the cloud system.
The 30 Seconds Sit to Stand - TEST RETEST (clinical setting) | 7 days after day 1
  In the clinical setting, the clinician asks the patient to sit in the middle of the chair, with the back straight, feet apart resting on the floor and in line with the shoulders. The patient has to rise from a sitting to a standing position as many times as possible in 30 seconds. With the results of this test, it is possible to evaluate a wide variety of skill levels, with scores ranging from 0 (for those unable to complete one repetition) to more than 20 repetitions (for the most physically fit individuals). For the automated test, the patient will wear a chest strap fixing the mobile phone over the sternum. On a sitting position, the patient will open the mHealth App and through the use of audible feedback, will receive the same test instructions as in the clinic. With the use of algorithms, the mHealth App will automatically count the total sit to stand repetitions within a 30 seconds period. After the test is completed, the data will be automatically sent to the cloud system.
The 30 Seconds Sit to Stand - DIURNAL CHANGE (home setting) | Day 1, day 3, and day 5 (within a week Mon, Wed, Fri)
  At home, for the automated test, the patient will wear a chest strap fixing the mobile phone over the sternum. On a sitting position, the patient will open the mHealth App and through the use of audible feedback, will receive the same test instructions as in the clinic. With the use of algorithms, the mHealth App will automatically count the total sit to stand repetitions within a 30 seconds period. After the test is completed, the data will be automatically sent to the cloud system.
The 20-meter Walk - TEST RETEST (clinical setting) | Day 1
  This test assesses gait speed and changes in patient's physical function over time. The clinician asks the patient to walk at a comfortable pace in a 20-meter unobstructed course and measures the time to perform the test. For the automated test, the patient will wear a chest strap fixing the mobile phone over the sternum. On a standing position, the patient will open the mHealth App and through the use of audible feedback, will receive the same test instructions as in the clinic. With the use of algorithms, the mHealth App will automatically determine when the 20-meter distance is reached and will say to the patient to gradually stop, measuring the total time to complete the test. After the test is completed, the data will be automatically sent to the cloud system.
The 20-meter Walk - TEST RETEST (clinical setting) | 7 days after day 1
  This test assesses gait speed and changes in patient's physical function over time. The clinician asks the patient to walk at a comfortable pace in a 20-meter unobstructed course and measures the time to perform the test. For the automated test, the patient will wear a chest strap fixing the mobile phone over the sternum. On a standing position, the patient will open the mHealth App and through the use of audible feedback, will receive the same test instructions as in the clinic. With the use of algorithms, the mHealth App will automatically determine when the 20-meter distance is reached and will say to the patient to gradually stop, measuring the total time to complete the test. After the test is completed, the data will be automatically sent to the cloud system.
The 20-meter Walk - DIURNAL CHANGE (home setting) | Day 1, day 3, and day 5 (within a week Mon, Wed, Fri)
  At home, for the automated test, the patient will wear a chest strap fixing the mobile phone over the sternum. On a standing position, the patient will open the mHealth App and through the use of audible feedback, will receive the same test instructions as in the clinic. With the use of algorithms, the mHealth App will automatically determine when the 20-meter distance is reached and will say to the patient to gradually stop, measuring the total time to complete the test. After the test is completed, the data will be automatically sent to the cloud system.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas O Dantas, PT, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil